CLINICAL TRIAL: NCT01014013
Title: A Prospective, Multicenter, Partially-Blinded, Randomized, Comparative Study to Evaluate the Safety, Tolerability and Efficacy of INVANZ Versus Ceftriaxone Sodium in the Treatment of Complicated Urinary Tract Infections in Adults
Brief Title: Safety and Tolerability of Ertapenem Sodium in the Treatment of Complicated Urinary Tract Infections (0826-055)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0826-055; MK0826-055; 2009_690
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Results first posted 2010-03-01 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ertapenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ertapenem sodium (MK0826) (Experimental): ertapenem sodium
  Interventions: Drug: ertapenem sodium (MK0826)
- ceftriaxone sodium (Active Comparator): ceftriaxone sodium
  Interventions: Drug: Comparator: ceftriaxone sodium

INTERVENTIONS:
Drug: ertapenem sodium (MK0826) — a single daily dose of ertapenem sodium 1.0g IV infused over 30 minutes, for 7-14 days (patients may be switched to oral ciprofloxacin after 3 doses of IV therapy if needed)
  Other Names: MK0826
  Arms: ertapenem sodium (MK0826)
Drug: Comparator: ceftriaxone sodium — a single daily dose of ceftriaxone 2.0g IV infused over 30 minutes, for 7-14 days (patients may be switched to oral ciprofloxacin after 3 doses of IV therapy)
  Arms: ceftriaxone sodium

SUMMARY:
The purpose of this study is to determine the efficacy of ertapenem sodium (Invanz) in treatment of complicated urinary tract infections with respect to the proportion of patients with a favorable microbiological response at 5-9 days post therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a suspected or documented complicated urinary tract infection
* Female patients must test negative for pregnancy and agree to use adequate birth control measures
* Nursing women must agree to defer breastfeeding until 5 days after completion of all study antibiotic therapy

Exclusion Criteria:

* Patients with complete obstruction of any portion of the urinary tract
* Patients with rapidly progressive or terminal illness
* Renal transplant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Park DW, Peck KR, Chung MH, Lee JS, Park YS, Kim HY, Lee MS, Kim JY, Yeom JS, Kim MJ. Comparison of ertapenem and ceftriaxone therapy for acute pyelonephritis and other complicated urinary tract infections in Korean adults: a randomized, double-blind, multicenter trial. J Korean Med Sci. 2012 May;27(5):476-83. doi: 10.3346/jkms.2012.27.5.476. Epub 2012 Apr 25. PMID 22563210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 9 Medical Centers of Korea between April 2008 and January 2009.
  Last patient has visited on 27 Feb 2009.
Pre-assignment Details: 1 patient was excluded due to ineligibility. The patient had a positive at screening pregnancy test.
Groups:
- MK0826: A single daily dose of MK0826 1.0 g intravenous infused over 30 minutes, for 7-14 days (patients may be switched to oral ciprofloxacin at a dose of 500 mg twice daily after 3 doses of parentheral therapy)
- Ceftriaxone: A single daily dose of 2.0 g Ceftriaxone sodium intravenous infused over 30 minutes, for 7-14 days (patients may be switched to oral ciprofloxacin at a dose of 500 mg twice daily after 3 doses of parentheral therapy)
Period: Overall Study
Arm/Group | MK0826 | Ceftriaxone
Started | 135 | 136
Adverse Event Reporting | 132 (Patients who received at least 1 dose of MK0826 parenteral therapy) | 135 (Patients who received at least 1 dose of Ceftriaxone parenteral therapy)
Completed Parenteral Therapy | 87 (Patients completing MK0826 as a single daily dose of 1.0g intravenous infusion at least 3 days) | 88 (Patients completing Ceftriaxone as a single daily dose of 2.0g intravenous infusion at least 3 days)
Completed | 84 (Patients who completed 7 days therapy including minimum 3 days of MK0826 parentheral therapy) | 80 (Patients who completed 7 days therapy including minimum 3 days of Ceftriaxone parentheral therapy)
Not Completed | 51 | 56
Not completed — Inclusion/Exclusion criteria not met | 1 | 3
Not completed — Clinical adverse experience | 4 | 2
Not completed — Laboratory adverse experience | 1 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Clinical/microbiologic failure | 1 | 2
Not completed — Pathogen culture = no growth | 26 | 34
Not completed — Negative urine culture | 2 | 0
Not completed — Pathogen resistant | 7 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Another antibiotic therapy required | 0 | 1
Not completed — Appendectomy | 1 | 0
Not completed — Inappropriate therapy duration, < 7 Days | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0826 | Ceftriaxone | Total
Number analyzed (Participants) | 135 | 136 | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (19.5) | 56.5 (17.6) | 55.9 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 126 | 245
  Male | 16 | 10 | 26
Stratum [Number; unit: participants] — Patients have enrolled who have complicated urinary tract infection with or without acute pyelonephritis
  participants
    Acute pyelonephritis | 103 | 107 | 210
    Other complicated urinary tract infection | 32 | 29 | 61
Duration of Symptoms(Days) [Mean (Standard Deviation); unit: Days] — The duration of clinical symptoms prior to study entry
  Days | 4.1 (4.6) | 4.7 (6.4) | 4.4 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Microbiological Response Assessment Profile
Description: The difference in favorable microbiological response rates between the 2 treatment groups (MK0826 response rate minus ceftriaxone response rate) was assessed
Time Frame: 5 to 9 days post-therapy
Population: Primary efficacy analysis was done for 137 evaluable patients (66 patients from MK0826 and 71 patients from Ceftriaxone)
Measure: Number; unit: Participants
Groups:
- MK0826: MK0826 as a single daily dose of 1.0 g intravenous infusion and be switched to oral ciprofloxacin at a dose of 500 mg twice daily and patients who 1) received a proper course of therapy. 2) had a confirmed diagnosis of complicated urinary tract infection, including acute pyelonephritis, 3) had not comment an major protocol violations, and 4) were microbiologically evaluable at the early follow-up (5 to 9 days post-therapy). Those patients were considered as evaluable.
- Ceftriaxone: Ceftriaxone sodium as a single daily dose of 2.0 g intravenous infusion and be switched to oral ciprofloxacin at a dose of 500 mg twice daily and patients who 1) received a proper course of therapy. 2) had a confirmed diagnosis of complicated urinary tract infection, including acute pyelonephritis, 3) had not comment an major protocol violations, and 4) were microbiologically evaluable at the early follow-up(5 to 9 days post-therapy) were considered as evaluable.(66 patients from MK0826 and 71 patients from Ceftriaxone). Those patients were considered as evaluable.
Arm/Group | MK0826 | Ceftriaxone
Number analyzed (Participants) | 66 | 71
Participants | 58 | 63
Statistical Analysis 1: Comparison: MK0826 vs Ceftriaxone; Test type: Non-Inferiority or Equivalence — The primary efficacy endpoint was based on the proportion of patients who had a favorable microbiological response assessment at follow-up 5 to 9 days post-therapy visit. The definition of non-inferiority is that the 95%(two-sided) confidence interval for the difference in response rate between the 2 treatment groups(MK0826 minus control group) contains zero and the lower limit of the CI is not less than -20 percentage points; the difference between two response rate = -0.8, 95% CI [-11.7 to 10.2], Standard Deviation 10.9

2. Primary Outcome: The Number of Patients Who Experience Any Drug-related Adverse Experiences Leading to Discontinuation of Parenteral Study Drug and the Number of Patients With Any Drug-related Serious Adverse Experiences (AEs) During Parenteral Treatment
Description: Safety was assessed by statistical and/or clinical review of all safety parameters, including adverse experiences, physical examination, vital signs, and laboratory results during parenteral therapy. As per the primary safety hypothesis, it was expected that, at the end of the parenteral therapy only, MK0826 would be similar to ceftriaxone with respect to the proportion of patients with any drug-related clinical or laboratory adverse experiences leading to discontinuation of study drug and also with respect to the proportion of patients with any serious drug-related adverse experiences.
Time Frame: Adverse experiences that occurred during the study parenteral therapy period were analyzed. The period of parenteral therapy is from 3 days up to 14 days
Population: Safety Analysis has been done 267 patients who received at least 1 dose of parenteral therapy (132 patients from MK0826 and 135 patients from Ceftriaxone)
Measure: Number; unit: Participants
Groups:
- MK0826: MK0826 as a single daily dose of 1.0 g intravenous infusion and be switched to oral ciprofloxacin at a dose of 500 mg twice daily and patients who received at least 1 dose of parentheral therapy
- Ceftriaxone: Ceftriaxone sodium as a single daily dose of 2.0 g intravenous infusion and be switched to oral ciprofloxacin at a dose of 500 mg twice daily and patients who received at least 1 dose of parentheral therapy
Arm/Group | MK0826 | Ceftriaxone
Number analyzed (Participants) | 132 | 135
Participants
  Discontinued due to drug-related clinical AEs | 1 | 0
  Serious drug-related clinical AEs | 0 | 0
  Discontinued due to drug-related laboratory AEs | 1 | 1
  Serious drug-related Laboratory AEs | 0 | 0

3. Secondary Outcome: Clinical Response Assessment Profile
Description: The difference in favorable clinical response rates between the 2 treatment groups (MK0826 response rate minus ceftriaxone response rate) was assessed
Time Frame: 5 to 9 days post-therapy
Population: Secondary efficacy analysis was done for 137 evaluable patients (66 patients from MK0826 and 71 patients from Ceftriaxone)
Measure: Number; unit: Participants
Arm/Group | MK0826 | Ceftriaxone
Number analyzed (Participants) | 66 | 71
Participants | 64 | 70
Statistical Analysis 1: Comparison: MK0826 vs Ceftriaxone; Test type: Non-Inferiority or Equivalence — The secondary efficacy endpoint was based on the proportion of patients who had a favorable clinical response assessment at follow-up 5 to 9 days post-therapy visit. The definition of non-inferiority is that the 95%(two-sided) confidence interval for the difference in response rate between the 2 treatment groups(MK0826 minus control group) contains zero and the lower limit of the CI is not less than -20 percentage points; the difference between two response rate = -1.7, 95% CI [-6.6 to 3.2], Standard Error of Mean 4.9

ADVERSE EVENTS:
Time Frame: Adverse experiences were recorded during parenteral therapy and for 14 days after the end of study therapy including oral study therapy (safety follow-up period)
Description: Safety was assessed by statistical and/or clinical review of all safety parameters, including adverse experiences (AE), physical examination, vital signs, and laboratory results
Arm/Group | MK0826 | Ceftriaxone
Serious Adverse Events (participants affected / at risk) | 12/132 | 8/135
Other Adverse Events (participants affected / at risk) | 85/132 | 90/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0826 (N=132) | Ceftriaxone (N=135)
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Renal abcess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders (Renal and urinary disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac discomfort (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Renal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0826 (N=132) | Ceftriaxone (N=135)
Diarrhea (Gastrointestinal disorders) | 27 | 20
Dyspepsia (Gastrointestinal disorders) | 8 | 15
Constipation (Gastrointestinal disorders) | 9 | 9
Nausea (Gastrointestinal disorders) | 8 | 9
Abdominal pain (Gastrointestinal disorders) | 4 | 8
Abdominal discomfort (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Epigastric discomfort (Gastrointestinal disorders) | 1 | 2
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastritis atrophic (Gastrointestinal disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 2
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 22 | 19
Dizziness (Nervous system disorders) | 2 | 4
Paraesthesia (Nervous system disorders) | 0 | 2
Burning sensation (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 3
Pyrexia (General disorders) | 3 | 1
Application site pain (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Face oedema (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Injection site erythema (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Injection site phlebitis (General disorders) | 0 | 1
Tenderness (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Herpes simplex (Infections and infestations) | 3 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Actinomycosis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 1
Urogenital trichomoniasis (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 10 | 8
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3
Cold sweat (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Blood pressure (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 3
Phlebitis (Vascular disorders) | 1 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
Hydroureter (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Gallbladder polyp (Hepatobiliary disorders) | 1 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 3 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 1
Conjunctivochalasis (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 4
Blood albumin decreased (Investigations) | 1 | 1
Blood potassium decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 2 | 0
Blood urea increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.